CLINICAL TRIAL: NCT04264910
Title: CALM Pregnancy: Feasibility of Mindfulness-based Prenatal Stress Reduction Using a Smart Phone Meditation Application
Brief Title: CALM Pregnancy: Feasibility of Calm for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Collaborators: Valley Perinatal Services (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: STUDY00010467
Record Dates: First submitted 2020-01-13; First posted 2020-02-11 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: Pregnant Women

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Calm Meditation (Experimental): Participants (n=49) will be provided free access to and asked to register for the consumer-based mobile meditation app on their phone. Participants (n=49) will then receive an email containing 28 weeks of free access to Calm. Participants (n=49) will be asked to use Calm at least 10 minutes per day and encouraged to use it as much as they would like during the intervention. This prescription mimics how a new, paying member would use the app (full exposure with autonomy).
  Interventions: Behavioral: Calm App
- Control (No Intervention): The control group will be asked to maintain normal activity and refrain from using Calm meditation app.

INTERVENTIONS:
Behavioral: Calm App — Calm is a subscription-based meditation app which provides guided meditations, sleep stories, soundscapes and calming music. Calm offers 7 Days of Calm for those new to meditation, the daily Calm, a meditation posted daily and a library of unique 10-12 minute meditations with topics related to acceptance, anxiety, self-compassion, and physical pain (to name a few).
  Arms: Calm Meditation

SUMMARY:
The purpose of this study is to determine the feasibility of using a consumer-based mindfulness app, Calm, to reduce stress during pregnancy. Women will be randomly assigned to an intervention group (i.e., Calm) or standard care group and asked to participate in at least 10 minutes of daily meditation for the duration of their pregnancy (i.e., 12-weeks' gestation up to date of birth).

Aim #1: Determine the feasibility (acceptability and demand) of using the Calm app at least 10-minutes per day for the duration of pregnancy (i.e., 12-weeks' gestation up to date of birth). Acceptability will be measured with an investigator-developed satisfaction survey.

Demand will be measured using time spent in meditation and meditations used (tracked by Calm).

For the intervention group, the benchmarks will be as follows:

1. Acceptability (i.e., satisfaction) 70% (n=34) of participants will report a 75% satisfaction,
2. Demand (i.e., time spent in meditation and meditations used,) 70% (n=34) of participants will adhere to ≥75% of prescribed meditation using Calm.

Aim #2: Determine the preliminary effects of using Calm at least 10-minutes per day for the duration of pregnancy (i.e., 12-16 weeks' gestation to date of birth) on stress. Stress will be measured using the Perceived Stress Scale (PSS) at baseline (i.e., 12-16-weeks' gestation) and every four weeks for the duration of the intervention using Ecological Momentary Assessment (i.e., text message). Stress will also be measured using cortisol serum at baseline (i.e., 12-16-weeks' gestation), and 32 weeks' gestation.

Exploratory Aim #3: The investigators will explore the preliminary effects of using Calm at least 10-minutes per day for the duration of pregnancy (i.e., 12-16 weeks' gestation to date of birth) on gestational age of birth, fetal weight, APGAR scores (i.e., health score), and neonatal complications with time spent in neonatal intensive unit (if applicable).

DETAILED DESCRIPTION:
Enrollment: Interested participants at Valley Perinatal Clinics will be asked for their email and will be sent a link to a brief (5-10 minute) eligibility screener via RedCap (See Eligibility screener). Eligible participants will be asked to watch a brief intake video followed by a 3-question quiz and asked to sign an electronic informed consent prior to completing any further surveys. After informed consents have been completed, participants (N=97) will be identified. Participants will be asked to complete a baseline questionnaire (See Surveys and Questionnaires document) and complete a medical history form, which will ask participants to include a history of medications. They also will be asked to sign a medical release form for their obstetrician. Ineligible participants will be notified by email according to the script (See Email Scripts document).

Randomization: Participants will be randomized into either the intervention (Calm App) or standard prenatal care control and given further instructions to begin participating (See Welcome Email in Email Scripts document).

Inclusion criteria are: (1) women 12-16 weeks pregnant, (2) >18 years of age, (3) English speaking, (3) not currently on steroid therapy, (4) willing to download the Calm app to their smartphone, and (5) have not practiced meditation or mindful movement more than 60 minutes a month in the past six months (6) willing to be randomized to one of two groups.

Control: The control group will be asked to maintain normal activity and refrain from using Calm meditation app.

Intervention: Participants (n=49) will be provided free access to and asked to register for the consumer-based mobile meditation app on their phone. Participants (n=49) will then receive an email containing 28 weeks of free access to Calm. Participants (n=49) will be asked to use Calm at least 10 minutes per day and encouraged to use it as much as they would like during the intervention. This prescription mimics how a new, paying member would use the app (full exposure with autonomy).

Meditation Tracking: Intervention participants (n=49) usage will be continuously tracked throughout the intervention by Calm.

Assessments: Intervention group participants will receive self-report questionnaires (via RedCap) at baseline, and post intervention only after informed consent has been is obtained. Included within these questionnaires the investigators will measure demographics (baseline only) and stress (using the Perceived Stress Scale), mindfulness (using the Mindfulness Attention Awareness Scale), depression (using the Edinburgh Postnatal Depression Scale), anxiety (using the Pregnancy Related Anxiety Questionnaire), self-compassion (using the Self-Compassion Scale), emotional regulation (using the Difficulties in Emotional Regulations Scale), gratitude (using the Gratitude During Pregnancy Scale), and childbirth experience (using the Childbirth Experience Questionnaire). Every four weeks for the duration of the intervention, the investigators will measure stress and mindfulness using Ecological Momentary Assessment (i.e., text message). At baseline, mid-intervention (24-26 weeks' gestation), and baseline (32-34 weeks' gestations) depression, anxiety, self-compassion, emotional regulation, and gratitude will be measured. After the baby is born, depression, anxiety, self-compassion, emotional regulation, and childbirth experience will be measured.

Stress will also be measured using cortisol serum at baseline (i.e., 12-16-weeks' gestation) and 32 weeks. These tests will be performed at no additional cost to the participant. The blood draws will be completed at Valley Perinatal Clinic by a trained employee of Valley Perinatal Clinic. No more than one tube (10 mL) of blood will be taken for the cortisol serum test.

A weekly log (via RedCap) recording any changes in medications will be sent to participants. Any changes in medications, specifically ISSRs, will be accounted for in data analysis.

Acceptability is dually defined as participant satisfaction with content (i.e., Calm) and perceived appropriateness and usefulness of the behavioral components (i.e., reminders, self-monitoring) for self-management. Acceptability will be measured with an investigator-developed satisfaction survey, included within the post intervention questionnaire. Acceptability will be defined as 70% (n=34) of participants reporting a 75% satisfaction.

Demand will be measured by compliance to the >10 mins/day and sustained use during pregnancy. Demand (i.e., time spent in meditation and meditations used) will be defined as 70% (n=34) of participants adhering to ≥75% of prescribed meditation using Calm. Demand will be measured by Calm (internally) and shared with Arizona State University.

ELIGIBILITY:
Inclusion Criteria:

* women 12-16 weeks pregnant
* 18 years of age
* English speaking
* not currently on steroid therapy
* willing to download the Calm app to their smartphone,
* have not practiced meditation or mindful movement more than 60 minutes a month in the past six months
* willing to be randomized to one of two groups.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — They have to be women
Enrollment: 97 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
Feasibility: Acceptability | Two weeks after delivery of baby
  Acceptability will be measured with an investigator developed survey
Feasibility: Demand (Time spent in meditation and meditations used) | At birth/delivery
  Demand will be gathered using meditation app usage data and defined as at least 70% of intervention group will adhere to at 75% of prescribed meditation

SECONDARY OUTCOMES:
Perceived Stress of Participant | baseline, 16, 20, 24, 28, 32, and 36 weeks' gestation, two weeks after delivery of baby
  Stress will be measured with PSS; scores may range from 0-40. Higher scores indicate higher stress levels.

OTHER OUTCOMES:
Age of Birth | At delivery
  Measured by gestational age
Fetal Weight | At delivery
  Measured by weight at birth
APGAR score | At delivery
  Baby's heart rate, muscle tone, and other vitals
Neonatal Complication | birth to one month of age
  Any complications post birth

CONTACTS AND LOCATIONS:
Locations (1):
- Arizona Biomedical Collaborative, Phoenix, Arizona, United States

IPD SHARING:
Plan to Share IPD: No